CLINICAL TRIAL: NCT07353099
Title: A Post-Authorization Safety Study (PASS) to Further Evaluate Real-World Safety in Patients With Congenital Thrombotic Thrombocytopenic Purpura (cTTP) Treated With Adzynma
Brief Title: A Study in Children and, Adults With Congenital Thrombotic Thrombocytopenic Purpura (cTTP) Treated With Adzynma
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-755-4007; EUPAS1000000870 (Other: EU PAS)
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
Keywords: Drug Therapy
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Data of participants who have received Adzynma for the treatment of cTTP will be collected retrospectively from medical records for approximately 5 years.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
Congenital thrombotic thrombocytopenic purpura (cTTP) is a rare blood disorder that some people are born with. It is caused by a problem in a gene passed down from parents to children, which affects the body's ability to produce a enzyme called ADAMTS13. This enzyme helps to cut down a larger form of protein called von Willebrand Factor (VWF). People with cTTP have low levels of ADAMTS13. Without ADAMTS13, large forms of vWF build up and cause blood clots in small blood vessels. These clots can block blood flow to vital organs, causing serious health problems. Adzynma is a human ADAMTS13 protein made in the laboratory. It works the same way as natural ADAMTS13 does and may provide higher levels of ADAMTS13.

The main aim of this study is to learn more about the risk of children and adults with cTTP treated with Adzynma developing antibodies that prevent Adzynma from working properly (called neutralizing antibodies) within 6 months after the first treatment and to understand the risk of allergic reactions within 7 days of the first treatment with Adzynma. Other aims are to better understand how safe treatment with Adzynma is over a longer period of time (called long-term safety) in children and adults with cTTP and to gather information about pregnancies and babies of women who have received Adzynma while pregnant.

Only data already available in the medical records of the people who received Adzynma for the treatment of cTTP in normal clinical practice will be reviewed and collected during this study.

ELIGIBILITY:
Inclusion criteria:

1. Is diagnosed with cTTP.
2. Had received commercially available Adzynma treatment for cTTP within the eligibility period of which there must be a recorded date and dose of at least one Adzynma administration in their medical chart.
3. Provides a signed informed consent form (informed consent form [ICF]; or assent and consent forms, if applicable), in accordance with local ethical and institutional requirements.

Exclusion criteria:

1. Has a history or presence of a functional ADAMTS13 inhibitor (that is, neutralizing antibodies to ADAMTS13/rADAMTS13).
2. Has concurrent use of an investigational drug or is enrolled in another clinical trial at the time of index Adzynma infusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult participants who have received Adzynma for the treatment of cTTP, either prophylactically or as on-demand therapy for acute episodes-including those who became pregnant during Adzynma treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Hypersensitivity Reactions Following the Index Adzynma Infusions | Up to 6 months following the index Adzynma infusion
  Index infusion is defined as the first Adzynma infusion date recorded in the medical record using commercially available Adzynma (excluding doses received in clinical studies or early access program).
Number of Participants With Neutralizing Antibodies to ADAMTS13 Following the Index Adzynma Infusions | Up to 6 months following the index Adzynma infusion
  Number of participants with neutralizing antibodies to ADAMTS13 following the index Adzynma infusions will be reported.

SECONDARY OUTCOMES:
Number of Participants With Long Term Safety Risk of Hypersensitivity Reactions Following the Index Adzynma Infusion | Up to 6 months of follow-up time from the index Adzynma infusion
  Number of participants with long term safety risk of hypersensitivity reactions following the index Adzynma infusion will be reported.
Number of Participants With Risk of Hypersensitivity Reactions After Each Administration of Adzynma Following the Index Infusion | Up to 7 days after each administration of Adzynma
  Number of participants with risk of hypersensitivity reactions after each administration of Adzynma following the index infusion will be reported.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From start of the study drug administration up to 5.5 years
  TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.
Gestational age at the Time of Infant Birth | At birth
  Gestational age at the time of infant birth will be reported.
Number of Participants With Spontaneous Abortion | Up to 5.5 years
  Spontaneous abortion is defined as pregnancy loss before 20 weeks of gestation.
Number of Participants With Stillbirth | Up to 5.5 years
  Stillbirth is defined as a fetal death after 20 weeks of gestation.
Number of Participants With Induced Abortion | Up to 5.5 years
  Number of participants with induced abortion will be reported.
Number of Participants With Live Birth | Up to 5.5 years
  Number of participants with live birth will be reported.
Number of Participants With any Pregnancy Related Complications | Up to 5.5 years
  Number of participants with any pregnancy related complications will be reported.
Number of Participants Categorized According to Gestational age of Greater Than or Equal to (>=) 37 Gestational Weeks and Less Than (<) 37 Gestational Weeks at Birth | At birth
  Number of participants categorized according to gestational age of greater than or equal to (>=) 37 gestational weeks and less than (<) 37 gestational weeks at birth will be reported.
Number of Infants Categorized According to Year of Birth | Up to 5.5 years
  Number of infants categorized according to year of birth will be reported.
Number of Infants With Normal Birth Weight | Up to 5.5 years
  Number of infants with normal birth weight will be reported.
Number of Infants With Small for Gestational Age (SGA) | Up to 5.5 years
  Small for gestational age is defined as birth size (weight, length or head circumference) less than the 10th centile for sex and gestational age.
Number of Infants With Congenital Anomaly Detected at the Time of Birth | At birth
  Number of infants with congenital anomaly detected at the time of birth will be reported.
Number of Participants by Breastfeeding Status While Receiving Adzynma | Up to 5.5 years
  Breastfeeding status during Adzynma treatment will be assessed and categorized based on response (Yes, No, or Unknown).
Number of Infant Categorized by Growth and Development Outcomes | Up to 5.5 years
  Number of infants categorized by growth and development outcomes (normal, abnormal [specify], or unknown) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/